CLINICAL TRIAL: NCT02996331
Title: Preventing Pressure Ulcers With Repositioning Frequency and Precipitating Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PRO00069413; 1R01NR016001-01A1 (NIH)
Record Dates: First submitted 2016-10-06; First posted 2016-12-19 (Estimated); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Pressure Ulcer
Keywords: Ulcer; Pressure Ulcer; Pathologic Processes; Skin Ulcer; Skin Diseases
MeSH Terms: conditions — Pressure Ulcer; Ulcer; Pathologic Processes; Skin Ulcer; Skin Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 2 hour arm (Active Comparator): All participants in this arm are assigned a 2-hour repositioning interval.
  Interventions: Other: 2 hour repositioning
- 3 hour arm (Experimental): All participants in this arm are assigned a 3-hour repositioning interval.
  Interventions: Other: 3 hour repositioning
- 4 hour arm (Experimental): All participants in this arm are assigned a 4-hour repositioning interval.
  Interventions: Other: 4 hour repositioning

INTERVENTIONS:
Other: 2 hour repositioning — Current PrU prevention protocols recommend repositioning moderate, high, and severe risk residents a minimum of every 2 hours. We propose to include low risk residents because studies suggest they too develop PrUs. New pressure redistribution mattresses may make 2 hour repositioning unnecessary, but optimal time between repositioning remains unclear. Aim is to determine differences in incidence of new PrUs in NH residents (low, moderate, high risk level) using VE surfaces and repositioned at 2, 3, and 4 hour frequencies.
  Arms: 2 hour arm
Other: 3 hour repositioning — It is expected that repositioning frequency can be extended for NH residents who are low, moderate, and high risk for pressure ulcer (PrU) development and on visco-elastic (VE) high-density foam support-surfaces without compromising PrU incidence. This intervention will include a 3 hour repositioning interval.
  Arms: 3 hour arm
Other: 4 hour repositioning — It is expected that repositioning frequency can be extended for NH residents who are low, moderate, and high risk for pressure ulcer (PrU) development and on visco-elastic (VE) high-density foam support-surfaces without compromising PrU incidence. This intervention will include a 4 hour repositioning interval.
  Arms: 4 hour arm

SUMMARY:
The purpose of this study is to determine whether repositioning frequency can be extended for nursing home (NH) residents who are low, moderate, and high risk for pressure ulcer (PrU) development. The investigators will also determine how changes in medical severity interact with changes in risk level and repositioning schedule to predict PrU development. This study will advance knowledge about repositioning frequency and clinically assessed PrU risk-level in relation to medical severity. Outcomes of this research will contribute to future guidelines for more precise preventive nursing practices and refinement of PrU prevention guidelines.

DETAILED DESCRIPTION:
The purpose of this 9 nursing homes (NH) cluster randomized study is to determine whether repositioning frequency can be extended for NH residents who are low, moderate, and high risk for pressure ulcer (PrU) development and on visco-elastic (VE) high-density foam support-surfaces without compromising PrU incidence. The investigators will also determine how changes in medical severity interact with changes in risk level and repositioning schedule to predict PrU development. PrUs result primarily from pressure over bony prominences that occlude blood flow to tissues. Current PrU prevention protocols recommend repositioning moderate, high, and severe risk residents a minimum of every 2 hours. The investigators propose to include low risk residents because studies suggest they too develop PrUs. New pressure redistribution mattresses may make 2 hour repositioning unnecessary, but optimal time between repositioning remains unclear. Aims are 1) determine differences in incidence of new PrUs in NH residents (low, moderate, high risk level) using VE surfaces and repositioned at 2, 3, and 4 hour frequencies; and 2) determine how medical severity components (measured by a modified Comprehensive Severity Index), changes in clinically assessed risk-level (low, moderate, high as measured by Braden Scale), repositioning schedule, and their interactions are associated with PrU development; and an Exploratory Aim: Evaluate PrU prevention intervention approach between NH groups repositioned at 2, 3, or 4 hour by: 1) comparing the intervention resource costs (VE surfaces, Leaf service/sensor use, fixed and variable labor costs for training and repositioning) and incremental cost-effectiveness ratio of cost per % reduction in PrUs, and 2) exploring staff and resident satisfaction with intervention approach. The investigators will randomly assign each NH to one of 3 study arms (2, 3, 4 hour) while providing standard nursing care. Leaf Patient Monitoring System will be used with sensor worn continuously to monitor repositioning. Periodic safety and care checks will be performed to ensure skin integrity. Residents admitted to study NHs for at least 3 days during the 6 week intervention, without an existing PrU, not using a specialty support surface, and of low, moderate, or high risk for PrU development will be included in analysis based on intention to treat. The outcome, no difference in PrU incidence, will determine whether repositioning frequency can be extended for low, moderate, high risk residents. Medical severity components and clinically assessed risk level will be examined for assessment to assessment change in relation to PrU development, thus identifying severity components associated with new PrUs. Data will be monitored by investigators daily. Data analysis and management will be performed by HSIR. NH staff and resident satisfaction with the intervention approach will be explored using focus groups. This study will advance knowledge about repositioning frequency and clinically assessed PrU risk-level in relation to medical severity. Outcomes of this research will contribute to future guidelines for more precise preventive nursing practices and refinement of PrU prevention guidelines.

ELIGIBILITY:
Inclusion Criteria:

* NH residents for a minimum of 3 days who use a VE-surface mattress, are without PrUs and are clinically assessed as low, moderate, or high risk for new PrU development will participate in their respective NH-wide repositioning frequency protocol.
* Participants will include residents at the time of study initiation and any newly admitted residents during the 6-week study period.

Exclusion Criteria:

* Newly admitted residents (less than 3 days)
* resident has been diagnosed with pre-existing pressure ulcer
* PrU Risk is severe (Braden score <= 9)
* the resident is cared for on a specialty bed (such as a bariatric bed)
* "do not turn" orders are present
* Allergy to adhesive

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2113 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-11 (Actual)

PRIMARY OUTCOMES:
Determine differences in PrU Incidence among NH in study arms. | 4 weeks
  Determine differences in the incidence of new PrUs in NH residents at low, moderate, and high risk using VE surfaces and repositioned at 2, 3, or 4 hour frequencies, in nine randomly assigned NHs over a 4-week period. We hypothesize that there will be no significant difference in PrU incidence between the 3 treatment arms in the study using three risk level groups: high risk (Braden Scale Score, 10-12), moderate risk (Braden Scale Score, 13-14), and low risk (Braden Scores >14). The hypothesis of no group-difference will be tested by examining whether the 95% confidence intervals of the rates of PrU and the 2-hour repositioning overlap. If they do, the hypothesis for no group-difference will be confirmed. Cumulative Incidence rate = [(# of residents with 1 or more new PrUs during intervention period) ÷ (# of residents participating in intervention for 3 or more days)] x 100; calculated for the full 4-week intervention period.

SECONDARY OUTCOMES:
Determine how medical severity components, changes in clinically assessed risk level, repositioning schedule, and their interactions are associated with development of PrUs. | 4 weeks
  Calculated severity score resulting from distillation of over 2,000 potential elements using the modified Comprehensive Severity Index (CSI) risk adjustment system. The more abnormal the signs/symptoms, the higher the severity score: Level 1 (normal to mild) - Level 4 (catastrophic, life-threatening, or likely to result in organ failure). PrU development will be examined and the PrU incidence rate will be modeled as a binary outcome. Additionally, generalized estimating equations (GEEs) will be used with model fit assessed using the quasi-likelihood information criterion (QIC). Robust standard errors, clustered at the facility level, will be employed to account for covariance among residents within facilities over time. To test the robustness of models, non-linear mixed models using PROC GLIMMIX will be employed as another option for modeling the data.
Evaluate cost-effectiveness of PrU prevention intervention approach between NH groups repositioned at 2, 3, or 4 hour intervals. | 4 weeks
  Comparing the intervention resource costs and incremental cost-effectiveness ratio of cost per % reduction in PrUs. Intervention cost will include labor cost, such as training time multiplied by wage & fringe rates of training participants and number of repositionings for each NH and study arm and time to conduct repositioning collected by Leaf system; multiplied by nurse wage & fringe rate. Non-labor cost inputs will include market prices paid fully depreciated over their respective useful life will be used to calculate daily equipment cost rates. Intervention cost by NH and study arm and incremental cost-effectiveness ratios (ICERs) will be calculated and compared for cost per % reduction in PrUs. Sensitivity analysis will be conducted with the range of observed repositioning times, nurse salaries, and market prices for non-labor inputs to assess the robustness of the ICERs and their sensitivity to labor and non-labor input prices.

CONTACTS AND LOCATIONS:
Overall Officials: Tracey Yap, PhD, RN, Principal Investigator — Duke University School of Nursing
Locations (1):
- Quinnipiac Valley Center, Wallingford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yap TL, Horn SD, Sharkey PD, Brooks KR, Kennerly S. The Nursing Home Severity Index and Application to Pressure Injury Risk: Measure Development and Validation Study. JMIR Aging. 2023 Feb 9;6:e43130. doi: 10.2196/43130. PMID 36757779
- [Derived] Yap TL, Alderden J, Sabol VK, Horn SD, Kennerly SM. Real-time Positioning Among Nursing Home Residents Living With Dementia: A Case Study. Wound Manag Prev. 2020 Jul;66(7):16-22. PMID 32614327
- [Derived] Sabol VK, Kennerly SM, Alderden J, Horn SD, Yap TL. Insight Into the Movement Behaviors of Nursing Home Residents Living With Obesity: A Report of Two Cases. Wound Manag Prev. 2020 May;66(5):18-29. PMID 32401731
- [Derived] Yap TL, Kennerly SM, Horn SD, Bergstrom N, Datta S, Colon-Emeric C. TEAM-UP for quality: a cluster randomized controlled trial protocol focused on preventing pressure ulcers through repositioning frequency and precipitating factors. BMC Geriatr. 2018 Feb 20;18(1):54. doi: 10.1186/s12877-018-0744-0. PMID 29463211